CLINICAL TRIAL: NCT01466530
Title: Effects of Preoperative Sublingual Misoprostol on Uterine Tone During Isoflurane Anaesthesia for Caesarean Section
Brief Title: Sublingual Misoprostol & Isoflurane During Caesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-2
Record Dates: First submitted 2011-10-27; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Pregnancy; Cesarean Delivery
Keywords: Full term pregnancy > 36 weeks; Cesarean delivery; General anesthesia
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): sublingual two moistened white coated placebo tablets
  Interventions: Drug: Placebo
- Misoprostol (Active Comparator): sublingual misoprostol (400 µg)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Placebo — received sublingual two moistened white coated placebo tablets which looked identical in size, colour, and packing to misoprostol tablet.
  Other Names: Group A
  Arms: Placebo
Drug: Misoprostol — sublingual misoprostol was given by putting two moistened tablets of misoprostol (400 µg) under the tongue and allowing them to dissolve (Misotac®, Sigma Pharmaceutical Industries, Egypt) (200 µg/tablet).
  Other Names: Group M
  Arms: Misoprostol

SUMMARY:
Misoprostol would reduce the uterine bleeding after caesarean delivery, without harmful effects on either mother or baby. The investigators postulated that the use of sublingual misoprostol during isoflurane anaesthesia for uncomplicated caesarean delivery would reduce maternal haemorrhage, uterine atonic effects, and the need for additional uterotonic agents, without harmful effects on either mother or baby. Therefore, the present study was designed to evaluate the effects of preoperative sublingual misoprostol on maternal blood loss, uterine tone, the need for additional oxytocin and neonatal outcome after elective caesarean delivery under isoflurane anaesthesia.

DETAILED DESCRIPTION:
Volatile anaesthetics including sevoflurane, desflurane, and isoflurane are often used during general anaesthesia for caesarean delivery. The cost effectiveness of isoflurane anaesthesia1 for caesarean delivery is widely used at many centres including the authors' centre, where general anaesthesia is commonly used for caesarean deliveries than did regional anaesthesia because of the refusal of many ladies for the later, especially in the light of evidence-based equivocal maternal or neonatal outcomes of both techniques. 2 However, isoflurane in similar to other inhalational anaesthetics have been shown a dose-dependent (from 0.5 to 2.35 minimum alveolar concentration (MAC)) induced myometrial relaxation in 25% of parturients with added risks of postpartum haemorrhage, 3-5 which may be mediated through the inhibition of the oxytocin-induced contraction,6 decrease in intracellular concentration of free calcium,7 inhibition of voltage-dependent calcium channels activity,8 and activation of adenosine triphosphate-sensitive potassium channels (K (ATP))9 of pregnant uterine smooth muscle.

Several uterotonics such as oxytocin reduce postpartum haemorrhage by inducing uterine contraction, but with added risks of haemodynamic adverse effects. 10 Sublingual or rectal misoprostol, a prostaglandin E1 analogue, in doses of 100 to 800 µg is safe and as effective as intravenous infusion of oxytocin in reducing blood loss and the need for additional oxytocin after caesarean delivery under either spinal or general anaesthesia, with occurrence of transient side effects such as nausea, shivering and pyrexia. 11-17 Misoprostol possess several advantages over oxytocin, including long shelf life, stability at room temperature, and possible buccal, rectal and sublingual administration. 11, 16The later has many advantages such as rapid uptake, long-lasting duration of effect, and greatest bioavailability, compared with other routes of misoprostol administration. 18 Up to our best knowledge, this trial was the first one studied the inhibitory effects of misoprostol on the uterine atonic effects of inhalational anaesthetics.

Based upon previous published data, 19 blood loss after caesarean delivery was normally distributed with standard deviation 560 ml. A priori power analysis indicated that 174 patients in each group would be sufficient to detect a 20% reduction in blood loss after caesarean delivery, with a type-I error of 0.05 and a power of 90%. The investigators added 10% more patients to account for patients dropping out during the study.

Patients were randomly allocated to receive sublingual 400 µg of misoprostol or identical placebo two tablets after tracheal intubation before surgery.

Anaesthetic management was standardized in all studied patients. Oral ranitidine 150 mg was given the night before and on the morning of surgery, with 0.3 mol/L sodium citrate (30 mL) given 15 min before induction. In the operating theatre women were positioned supine on the operating table with 15° firm rubber wedge under the right hip to effect left uterine displacement. A slow 500-mL i.v. infusion of lactated Ringer's solution was given to all subjects over 20 min.

Subjects were monitored with electrocardiography, non-invasive blood pressure, pulse oximetry (SpO2), and end-tidal carbon dioxide concentration (EtCO2). After pre-oxygenation for 5 min, rapid-sequence induction was performed with propofol 1.5-2 mg/kg followed by suxamethonium 1.5 mg/kg after loss of verbal response. Cricoid pressure was applied after loss of consciousness and was released after correct placement of the tracheal tube had been confirmed.

After tracheal intubation, subjects were allocated randomly to two groups by drawing sequentially numbered sealed opaque envelopes containing a software-generated randomisation code (Random Allocation Software, version 1.0.0, Isfahan University of Medical Sciences, Isfahan, Iran). The parturients in the placebo group (n = 183) received sublingual two moistened white coated placebo tablets which looked identical in size, colour, and packing to misoprostol tablet. In the misoprostol group (n = 183), sublingual misoprostol was given by putting two moistened tablets of misoprostol (400 µg) under the tongue and allowing them to dissolve (Misotac®, Sigma Pharmaceutical Industries, Egypt) (200 µg/tablet). The anaesthesiologists who gave the anaesthetics and study tablets were blinded to the study randomization and were not involved in collecting of the patients' data. All staff in the operating room were unaware of the randomization code.

Anaesthesia was maintained with 0.5-1 MAC of isoflurane with nitrous oxide 50% in oxygen to maintain the heart rate and blood pressure within 20% of baseline values. Neuromuscular block was maintained with vecuronium 0.06 mg/kg. The lungs were ventilated using a tidal volume of 8 mL/kg, an inspiration-expiration ratio of 1: 2, and at a respiratory rate necessary to maintain an EtCO2 of 30-35 mm Hg. An infusion of lactated Ringer's solution 800 mL was given to all subjects during the procedure. Induction to delivery (I-D) times was recorded using a stopwatch.

After the umbilical cord was clamped, a 10-unit infusion of oxytocin in 500 mL of 5% glucose was started. Intravenous midazolam 0.05 mg/kg and fentanyl 2.0 µg/kg were given and end-tidal concentration of the nitrous oxide was increased to 70%.

The obstetrician who was blinded to the study group, assessed the uterine tone by palpation every three minutes after delivery of the placenta and rated the degree of uterine contraction on a 10-cm VAS (0: well contracted; 10: completely relaxed). If uterine tone remained unsatisfactory after 3 min, an additional 5-unit bolus of oxytocin was administered.

All neonates were assessed by a paediatrician unaware of the randomisation code as regarding their Apgar scores at 1 and 5 min, arterial blood pressure, heart rate, temperature and arterial oxygen saturation.

At the end of surgery, isoflurane and nitrous oxide were discontinued, residual neuromuscular block was antagonised and the patients were extubated. Postoperative analgesia was achieved with morphine, tramadol and paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I and II
* parturients aged 18-35 years
* uncomplicated singleton pregnancies
* Gestational age >= 36 weeks
* elective caesarean delivery
* refused regional anaesthesia
* requested general anaesthesia.

Exclusion Criteria:

* allergy to prostaglandins
* bronchial asthma
* anaemia
* bleeding disorders
* cardiac diseases
* inflammatory bowel diseases
* multiple pregnancies
* preeclampsia
* placenta praevia
* abruptio placenta
* previous postpartum haemorrhage
* antepartum haemorrhage
* grand multiparity
* uterine fibroids
* intrauterine growth restriction
* fetal abnormality

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 366 (Actual)
Dates: Start 2006-01; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
estimated blood loss after caesarean delivery | up to 24 hours
  estimated blood loss (EBL) = pregnancy blood volume (ml) (EBV) x [preoperative haematocrit - postoperative haematocrit] / preoperative haematocrit, where EBV measured as shown in the following formula; (0.75 x {[maternal height (inches) x 50] + [maternal weight in pounds x 25]})

SECONDARY OUTCOMES:
uterine tone | 5 min, 10 min, 15 min, 20 min, 25 min, 30 min
  The obstetrician who was blinded to the study group, assessed the uterine tone by palpation every three minutes after delivery of the placenta and rated the degree of uterine contraction on a 10-cm VAS (0: well contracted; 10: completely relaxed).
need for additional oxytocin | 8 hrs
  If uterine tone remained unsatisfactory for 3 min after delivery, an additional 5-unit bolus of oxytocin was administered. The number of patients received oxytocin was recorded
haematocrit levels | 24 hours, 48 hours
  haematocrit levels was recorded before and 48 hours after cesarean delivery
neonatal outcome | 1 min and 5 min
  Apgar score and clinical signs after delivery
adverse effects | 48 hours
  the presence of postoperative side effects such as nausea and vomiting, diarrhoea, abdominal pain, pyrexia, and shivering were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Principal Investigator — College of medicine, Manoura University
Locations (1):
- College of Medicine, Mansoura University, Al Mansurah, DK, Egypt